CLINICAL TRIAL: NCT00970970
Title: Visualizing VEGF Producing Lesions in Von Hippel-Lindau Disease
Brief Title: Visualizing Vascular Endothelial Growth Factor (VEGF) Producing Lesions in Von Hippel-Lindau Disease
Acronym: VHLimage
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: VHL Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: METc2009.119
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Von Hippel-Lindau Disease; Hemangioblastoma; Renal Cell Carcinoma; Pheochromocytoma; Pancreatic Neuroendocrine Tumor
Keywords: Vascular endothelial growth factor; von Hippel Lindau disease; molecular imaging; biomarker
MeSH Terms: conditions — von Hippel-Lindau Disease; Hemangioblastoma; Carcinoma, Renal Cell; Pheochromocytoma; Adenoma, Islet Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be taken at day 1 and at the day of the MRI scan for analysis of VEGF pathway related biomarkers (such as plasma VEGF, PDGF, placental growth factor (PlGF), soluble VEGF receptors) and endothelial activation markers (such as Von Willebrand Factor (VWF), plasminogen activator inhibitor type 1 antigen (PAI-1), tissue-type plasminogen activator antigen (t-PA) and circulating endothelial cells (CECs)). DNA analysis for evaluation of polymorphisms in genes involved in angiogenesis is optional. In available biopsy or resection specimens, additional molecular staining of VEGF pathway related proteins will be performed (such as VEGF, VEGF receptors, HIF).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Von Hippel Lindau: Adult patients with Von Hippel-Lindau disease
  Interventions: Other: 89Zr bevacizumab PET scan

INTERVENTIONS:
Other: 89Zr bevacizumab PET scan — Patients will be injected intravenously with 37 MBq, protein dose 5 mg 89Zr-bevacizumab at day 0. PET scans will be done at day 4.
  Other Names: VEGF imaging

SUMMARY:
Von Hippel Lindau disease (VHLD) is an inherited syndrome characterized by vascular malformations, kidney cancer, adrenal gland and pancreas tumors. The VHL protein is not functional in the different disease associated lesions which results in production of high amounts of vascular endothelial growth factor (VEGF). Currently there are no clinical, radiographic or molecular markers that can predict the natural history of a given lesion. With 89Zr-bevacizumab positron emission tomography (PET) scanning, VEGF can be visualized and quantified.

The investigators hypothesize that 89Zr-bevacizumab PET imaging is a useful tool to predict the behaviour of disease associated lesions in patients with VHLD.

Adult patients with VHLD who have had routine magnetic resonance imaging (MRI) scans of central nervous system (CNS) and abdomen will undergo a 89Zr-bevacizumab PET scan. MRI will be repeated within 12 months.

ELIGIBILITY:
Inclusion Criteria:

* clinically or genetically proven VHLD
* at least 1 measurable, VHL associated lesion in the CNS
* routine MRI of the CNS ≤ 6 weeks before inclusion
* routine CT or MRI of upper abdomen ≤ 3 months before inclusion or planned ≤ 3 months after 89Zr-bevacizumab PET scan
* age ≥ 18 years
* written informed consent must be given according to good clinical practice (GCP), and local regulations

Exclusion Criteria:

* pregnancy
* any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol, those conditions should be discussed with the patient before registration in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from a tertiary referral center for Von Hippel-Lindau disease.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2009-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Detection rate of VHL associated lesions with 89Zr-bevacizumab PET scans in patients with VHLD | An 89Zr-bevacizumab PET scan will be performed within 6 weeks after routine MRI CNS investigation, MRI will be repeated within 12 months.

SECONDARY OUTCOMES:
Progressive lesions within 12 months, defined as new lesions or lesions that show an increase in size of at least 5% of the longest diameter on MRI, or lesions that become symptomatic | The baseline MRI scan will be compared with a follow-up MRI scan within 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sjoukje Oosting, MD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands